CLINICAL TRIAL: NCT05033262
Title: Adaptation of the OurCareWishes.Org ACP Platform for Persons With Dementia in NHs and Their Caregivers
Brief Title: Our Care Wishes - Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 834878; P30AG064105-01 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-09-02 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Dementia; Alzheimer Disease; Memory Impairment
Keywords: Advance Care Planning; Shared Decision-Making; Web-Based Platform; Memory Care; Nursing Homes
MeSH Terms: conditions — Dementia; Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants who are allocated to the control arm will complete baseline measures and then receive usual advanced care planning care and discussions with the nursing facility staff. Control arm participants will not review the Our Memory Care Wishes website. Participants will complete follow up measures one week after the baseline interview.
- Intervention (Experimental): Participants allocated to the intervention group will complete baseline measures. Then, the participant will review the Our Memory Care Wishes website and enter advanced care planning decisions and preferences into the website. Participants will complete follow up measures one week after the baseline interview. Participants receiving the intervention will complete additional follow up measures which include surveys measuring the ease of use of the website.
  Interventions: Other: Our Memory Care Wishes

INTERVENTIONS:
Other: Our Memory Care Wishes — Our Memory Care Wishes is a web-based advance care planning platform designed for persons living with dementia in nursing homes to discuss and document healthcare and daily life preferences with the help of shared decision-makers. Penn researchers meet via Zoom with PLWD and their SDMS and nursing home staff to facilitate website completion.
  Arms: Intervention

SUMMARY:
This Our Care Wishes- Dementia pilot study is adapting an existing successful online advance care planning platform to the specific needs of persons living with dementia and shared decision-makers (SDMs) and testing the usability and acceptability among nursing home residents and SDMs.

ELIGIBILITY:
Inclusion Criteria:

* Eligible PLWD will be receiving short-or long-term care at a participating NH, have documented moderate to severe cognitive impairment as measured by the Cognitive Function Scale included in the Minimum Data Set 3.0, 65 and have an identified SDM.

Exclusion Criteria:

* Participants are not eligible discharged from participating NHs, or do not have access to a telephone or video chat.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dyads (i.e., persons living with dementia (PLWD) and their shared decision-makers (SDMS) were initially recruited by nursing home staff. Then, study staff read an assent script to and reviewed study procedures with interested SDMs. SDMs who agreed to participate were sent a copy of the study summary and assent script. After verbal assent was acquired, dyads (PLWDs and SDMs) were assigned to the intervention group or control arm.
Pre-assignment Details: Enrolled participants are organized into 4 individual groups: PLWDs & SDMs in the intervention and control arms. Dyads in all study arms who stopped answering study team calls after initial verbal telephone consent and did not complete the baseline interview were not considered enrolled and are excluded from the "Baseline & Follow Up Surveys" period below.
  Demographics were collected during the baseline interview.
  Nursing home staff were not enrolled in the study.
Groups:
- PLWD: Control: Participants living with dementia randomized to the control group will receive usual advanced care planning help from nursing facility staff and will not complete the Our Memory Care Wishes website.
  Participants will complete surveys that capture confidence in decision-making at baseline and 1 week. Participants will complete these surveys alongside their shared decision makers.
- SDMs: Control: Shared decision-makers of persons living with dementia randomized to the control group will work with their care receiver to have usual advanced care planning discussions with nursing facility staff. SDMs in the control group will not complete the Our Memory Care Wishes website.
  SDMs will complete surveys that capture confidence in decision-making at baseline and 1 week. SDMs will complete these surveys alongside the nursing home resident they care for.
- PLWD: Intervention: Persons living with dementia (PLWD) randomized to the intervention group will complete a baseline interview alongside their shared decision-maker (SDM) that collects demographics and their confidence in decision-making.
  Then PLWDs will work with their SDM to complete the Our Memory Care Wishes website with the PLWD. Our Memory Care Wishes is a web-based advance care planning platform designed for persons living with dementia in nursing homes to discuss and document healthcare and daily life preferences with the help of shared decision-makers.
  1 week after completing the website, PLWDs will complete a follow up interview collecting their confidence in decision-making, ratings of the website and how COVID has affected their decision-making.
- SDMs: Intervention: Shared decision-makers (SDMs) of persons living with dementia (PLWD) randomized to the intervention group will complete a baseline interview that collects demographics and their confidence in decision-making when it comes to being a surrogate for the PLWD.
  Then, SDMs will complete the Our Memory Care Wishes website with the PLWD. Our Memory Care Wishes is a web-based advance care planning platform designed for persons living with dementia in nursing homes to discuss and document healthcare and daily life preferences with the help of shared decision-makers.
  1 week after completing the website, SDMs will complete a follow up interview collecting their confidence in decision-making, ratings of the website and how COVID has affected their decision-making.
Period: Overall Study
Arm/Group | PLWD: Control | SDMs: Control | PLWD: Intervention | SDMs: Intervention
Started (After initial verbal screening and randomization, 4 dyads did not participant in the study. These dyads stopped answering calls after initial verbal consent.) | 3 | 3 | 4 | 4
Completed | 2 | 3 | 4 | 3
Not Completed | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: PLWDs and their SDMs in control and intervention study arms met with study staff and nursing home staff to complete baseline interviews. At baseline, demographics and confidence levels in decision-making were collected for both SDMs and PLWDs.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLWD: Control | SDMs: Control | PLWD: Intervention | SDMs: Intervention | Total
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 2 | 3
  >=65 years | 3 | 2 | 4 | 2 | 11
Age, Continuous [Mean (Full Range); unit: years] | 78.6 [70 to 88] | 64 [40 to 80] | 89.3 [87 to 91] | 65.5 [53 to 83] | 74.8 [40 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 3 | 8
  Male | 2 | 1 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 2 | 2 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 3 | 3 | 10
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Adapted Decision Making Confidence Scale
Description: Items from the Surrogate Decision-Making Confidence Scale and 9-item ACP Engagement Survey were used and adapted to capture the confidence in advanced care planning decision-making from both persons living with dementia and their shared decision-maker' points of view. The scale utilizes a Likert scale with values ranging from 1 (not confident at all) to 5 (very confident).
Time Frame: Baseline
Population: SDMs and PLWDs in all study arms that completed the baseline interview were analyzed.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- PLWDs: Intervention: Persons living with dementia (PLWD) randomized to the intervention group will complete a baseline interview alongside their shared decision-maker (SDM) that collects demographics and their confidence in decision-making.
  Then PLWDs will work with their SDM to complete the Our Memory Care Wishes website with the PLWD. Our Memory Care Wishes is a web-based advance care planning platform designed for persons living with dementia in nursing homes to discuss and document healthcare and daily life preferences with the help of shared decision-makers.
  Our Memory Care Wishes: Our Memory Care Wishes is a web-based advance care planning platform designed for persons living with dementia in nursing homes to discuss and document healthcare and daily life preferences with the help of shared decision-makers. Penn researchers meet via Zoom with PLWD and their SDMS and nursing home staff to facilitate website completion.
Arm/Group | PLWD: Control | SDMs: Control | PLWDs: Intervention | SDMs: Intervention
Number analyzed (Participants) | 3 | 3 | 4 | 4
score on a scale | 4.8 [4.5 to 5] | 4.7 [4.2 to 5] | 3.7 [1 to 5] | 5 [5 to 5]

2. Primary Outcome: Post Adapted Decision Making Confidence Scale
Description: Items from the Surrogate Decision-Making Confidence Scale and 9-item ACP Engagement Survey were used and adapted to capture the confidence in advanced care planning decision-making from both persons living with dementia and their shared decision-maker' points of view. The scale utilizes a Likert scale with values ranging from 1 (not confident at all) to 5 (very confident). This is the second time point the measure was collected.
Time Frame: 1 week
Population: 1 PLWD from the control group and 1 SDM from the Intervention group were lost to follow up. Data was not collected at this timepoint and so were not analyzed.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | PLWD: Control | SDMs: Control | PLWD: Intervention | SDMs: Intervention
Number analyzed (Participants) | 2 | 3 | 4 | 3
units on a scale | 4.9 [4.8 to 5] | 4.7 [4.4 to 5] | 4.25 [2 to 5] | 5 [5 to 5]

3. Primary Outcome: Website Ease of Use
Description: This scale measures the ease of use of the website. This scale uses a Likert scale from 0 (very hard) to 10 (very easy). These data were collected from PLWDs and SDMs in the intervention group.
Time Frame: 1 week
Population: SDMs tended to navigate the website and use the website to facilitate advanced care planning discussions with PLWDs. PLWDs participated in conversations about advanced care planning decisions but often did not actively use the website and so were not always able to answer or understand the questions regarding the website. In the end, only one PLWD from the intervention group was able to answer the questions about the website's ease of use. Thus, the score below indicates that PLWD's rating.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- PLWD: Intervention: Persons living with dementia (PLWD) randomized to the intervention group will complete a baseline interview alongside their shared decision-maker (SDM) that collects demographics and their confidence in decision-making.
  Then PLWDs will work with their SDM to complete the Our Memory Care Wishes website with the PLWD. Our Memory Care Wishes is a web-based advance care planning platform designed for persons living with dementia in nursing homes to discuss and document healthcare and daily life preferences with the help of shared decision-makers.
Arm/Group | PLWD: Intervention | SDMs: Intervention
Number analyzed (Participants) | 1 | 3
score on a scale | 7 [7 to 7] | 9 [8 to 10]

4. Primary Outcome: Rate of ACP Website Completion - Time
Description: This tool measured total time spent by participants on the advance care planning website. Total time in minutes spent on the website were collected. Because SDMs navigated the website with the PLWD alongside them, this measure was only used to SDMs in the intervention group.
Time Frame: 1 week
Population: Total time SDMs spent navigating the Our Memory Care Wishes website was captured for each SDM in the intervention group.
Measure: Mean (Full Range); unit: minutes
Arm/Group | SDMs: Intervention
Number analyzed (Participants) | 4
minutes | 42.93 [35.25 to 78.75]

5. Primary Outcome: Rate of ACP Website Completion - Questions Completed
Description: This tool measured what percentage of the website was completed by participants. Because SDMs navigated the website with the PLWD alongside them, this measure was only associated with SDMs in the intervention group.
Time Frame: 1 week
Population: Percentage of website completed was captured for SDMs as they were primary navigators of the website.
Measure: Mean (Full Range); unit: percentage of website completed
Arm/Group | SDMs: Intervention
Number analyzed (Participants) | 4
percentage of website completed | 69 [21 to 92]

6. Other Pre Specified Outcome: COVID-19 Impact Questionnaire
Description: Participants were asked if their healthcare preferences changed due to the COVID-19 pandemic. Items included:
  1. Since COVID, planning for the future is: (1) less important (2) more important, or (3) the same
  2. Since COVID, the sense of urgency to name a supportive decision maker has: (1) increased (2) decreased, or (3) remained the same.
  3. Since COVID, my preferences for decisions about breathing machines (ventilators) have: (1) changed or (2) remained the same.
  4. Since COVID, my preferences for going to the hospital for care versus receiving treatment in place have:(1) changed, or (2) remained the same.
Time Frame: 1 week
Population: 1 PLWD in the control group was lost to follow up.
  1 SDM in the control group was lost to follow up.
  1 PLWD in the intervention group was lost to follow up.
  1 SMD in the intervention group was lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | PLWD: Control | SDMs: Control | PLWD: Intervention | SDMs: Intervention
Number analyzed (Participants) | 2 | 3 | 3 | 3
Participants
  Participants who reported a change in importance level for planning for the future since COVID-19. | 1 | 1 | 1 | 1
  Change in the sense of urgency to name a supportive decision maker since COVID-19 | 0 | 2 | 0 | 1
  Participants who reported a change in breathing machine preferences since COVID-19. | 0 | 1 | 0 | 1
  Participants whose preferences for going to the hospital for care versus receiving treatment changed | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 10 months
Description: 14 out of 14 participants analyzed. No adverse events occured.
Groups:
- Control: Participants randomized to the control group will receive usual advanced care planning help from nursing facility staff and will not complete the Our Memory Care Wishes website. Participants will complete surveys that capture confidence in decision-making at baseline and 1 week.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT05033262/Prot_SAP_000.pdf